CLINICAL TRIAL: NCT02153073
Title: Omega-3 Fatty Acid Ethyl Esters (Lotriga) Granular Capsules Special Drug Use Surveillance (Long-term Use Survey)
Brief Title: Evaluation of the Safety and Efficacy of Long-term Use of Omega-3 Fatty Acid Ethyl Esters
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 142-011; JapicCTI-142457 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Hyperlipidemia
Keywords: Pharmacological therapy
MeSH Terms: conditions — Hyperlipidemias | interventions — Omacor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Omega-3 fatty acid ethyl esters 2 g: Omega-3 fatty acid ethyl esters 2 g, administered orally once or twice daily after meals
  Interventions: Drug: Omega-3 fatty acid ethyl esters

INTERVENTIONS:
Drug: Omega-3 fatty acid ethyl esters — Omega-3 fatty acid ethyl esters granular capsules
  Other Names: Lotriga Granular Capsules

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term use of granular capsule formulation of omega-3 fatty acid ethyl esters (Lotriga Granular Capsules) in patients with hyperlipidemia in daily medical practice

DETAILED DESCRIPTION:
This special drug use surveillance on long-term use of granular capsule formulation of omega-3 fatty acid ethyl esters (Lotriga Granular Capsules) was designed to investigate the frequency of adverse events in patients with hyperlipidemia The usual adult dosage is 2 g of omega-3 fatty acid ethyl esters administered orally once daily after meals. However, the dosage can be increased up to twice daily (at a dose of 2 g) depending on the participant's triglyceride level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hyperlipidemia

Exclusion Criteria:

1. Patients with hemorrhage (e.g., hemophilia, capillary fragility, gastrointestinal ulcer, urinary tract hemorrhage, hemoptysis, or vitreous hemorrhage)
2. Patients with a history of hypersensitivity to ingredients in granular capsule formulation of omega-3 fatty acid ethyl esters

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hyperlipidemia
Sampling Method: Probability Sample
Enrollment: 3084 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 570 investigative sites in Japan, from 29 May 2013 to 31 May 2017.
Pre-assignment Details: Participants with a historical diagnosis of hyperlipidemia were enrolled. Participants received interventions as part of routine medical care.
Groups:
- Omega-3 Fatty Acid Ethyl Esters 2 g: Oral administration with granular capsule formulation of 2 g of omega-3 fatty acid ethyl esters once daily for 12 months. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Started | 3084
Completed | 2786
Not Completed | 298
Not completed — Case Report Forms Uncollected | 230
Not completed — Protocol Deviation | 68

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 2786
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1382
  Male | 1404
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 2786
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 2765
    Inpatient | 21
BMI [Mean (Standard Deviation); unit: Kilograms (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)/meter (m)^2
    number analyzed (Participants) | 1941
    (all) | 24.94 (4.097)
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Medical Complications | 566
    Had Presence of Medical Complications | 2220
Drinking Habits [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 687
    No | 1609
    Unknown | 490
Triglycerides (TG) in Fasted Condition [Milligrams (mg)/ Deciliter (dL)] [Count of Participants; unit: Participants]
  < 150 mg/dL | 298
  >= 150 mg/dL and < 400 mg/dL | 824
  >= 400 mg/dL and < 500mg/dL | 64
  >= 500 mg/dL and < 750mg/dL | 43
  >= 750mg/dL | 16
  Not Measured | 1541
TG in Non-Fasted Condition (mg/dL) [Count of Participants; unit: Participants]
  < 150 mg/dL | 287
  >= 150 mg/dL and < 400 mg/dL | 762
  >= 400 mg/dL and < 500mg/dL | 78
  >= 500 mg/dL and < 750mg/dL | 82
  >= 750mg/dL | 31
  Not Measured | 1546
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 1430
  Current Smoker | 307
  Ex-Smoker | 496
  Unknown | 553
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had No Predisposition to Hypersensitivity | 2520
    Had Predisposition to Hypersensitivity | 133
    Unknown | 133
Duration of Diagnosis of Hyperlipidemia [Mean (Standard Deviation); unit: Years] — Mean duration between start of study and first time of diagnosis of hyperlipidemia was reported. Population: Population Analysis Description: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 2074
    (all) | 3.13 (4.755)
Surgery within One Month before Dosing [Count of Participants; unit: Participants]
  Had No Surgery within One Month before Dosing | 2762
  Had Surgery within One Month before Dosing | 24
Pregnancy Status during the Administration Period [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 1382
    Not Pregnant | 1381
    Pregnant | 1

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline in Lipid Parameters - Triglycerides (TG)
Description: Percent change from baseline in TG values as one of lipid parameters in fasted condition at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. The analyzed numbers were participants who were evaluable for this outcome measure at the given time point.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 1018
Percent change | -20.54 (40.259)

2. Secondary Outcome: Percent Change From Baseline in Lipid Parameters - LDL Cholesterol (LDL-C)
Description: Percent change from baseline in LDL-C values as one of lipid parameters in fasted condition at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 469
Percent change | 7.73 (82.486)

3. Secondary Outcome: Percent Change From Baseline in Lipid Parameters - VLDL Cholesterol (VLDL-C)
Description: Percent change from baseline in VLDL-C values as one of lipid parameters in fasted condition at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.The analyzed numbers were participants who were evaluable for this outcome measure at the given time point.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 22
Percent change | -14.15 (57.833)

4. Secondary Outcome: Percent Change From Baseline in Lipid Parameters - Apo-B
Description: Percent change from baseline in Apo-B values as one of lipid parameters in fasted condition at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 35
Percent change | -7.21 (12.979)

5. Secondary Outcome: Percent Change From Baseline in Lipid Parameters - Apo-CIII
Description: Percent change from baseline in Apo-CIII values as one of lipid parameters in fasted condition at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 31
Percent change | -5.49 (23.117)

6. Secondary Outcome: Percent Change From Baseline in Lipid Parameters - Lipoprotein
Description: Percent change from baseline in Lipoprotein values as one of lipid parameters in fasted condition at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 28
Percent change | -2.98 (28.385)

7. Secondary Outcome: Percent Change From Baseline in Lipid Parameters -Remnant-Like Particles-Cholesterol (RLP-C)
Description: Percent change from baseline in RLP-C values as one of lipid parameters in fasted condition at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 39
Percent change | -22.42 (94.776)

8. Secondary Outcome: Percent Change From Baseline in Lipid Parameters - Total Cholesterol (TC)
Description: Percent change from baseline in TC values as one of lipid parameters at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 1327
Percent change | -4.26 (17.488)

9. Secondary Outcome: Percent Change From Baseline in Lipid Parameters - Non-HDL Cholesterol (Non-HDL-C)
Description: Percent change from baseline in Non-HDL-C values as one of lipid parameters at final assessment point (up to Month 12) was reported.
Time Frame: Baseline, up to 12 months (Final Assessment Point)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 51
Percent change | -1.42 (23.495)

10. Primary Outcome: Number of Participants Who Had One or More Adverse Events (AE) and Serious Adverse Events (SAE)
Time Frame: Up to Month 12
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 2786
Participants
  AE | 130
  SAE | 26

ADVERSE EVENTS:
Time Frame: Up to Month12
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
All-Cause Mortality (participants affected / at risk) | 10/2786
Serious Adverse Events (participants affected / at risk) | 26/2786
Other Adverse Events (participants affected / at risk) | 38/2786
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omega-3 Fatty Acid Ethyl Esters 2 g (N=2786)
Sinusitis (Infections and infestations) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Dementia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Deep vein thrombosis (Vascular disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Rectal prolapse (Gastrointestinal disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Drowning (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Road traffic accident (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omega-3 Fatty Acid Ethyl Esters 2 g (N=2786)
Diarrhoea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Hepatic function abnormal (Hepatobiliary disorders) | 7
Bronchitis (Infections and infestations) | 7
Viral upper respiratory tract infection (Infections and infestations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT02153073/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT02153073/SAP_001.pdf